CLINICAL TRIAL: NCT01296321
Title: Tailored Internet-administrated Treatment of Panic Symptoms - A Randomised Controlled Trial
Acronym: NOVA III
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Gerhard Andersson/Professor, Linköping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-FAS-2008-1145
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Anxiety Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Waiting Lists

ARMS (2):
- Tailored Internet-delivered CBT (Experimental): Behavioral: Tailored Internet-delivered CBT
  Interventions: Behavioral: Tailored Internet-administrated CBT-Treatment
- Waitlist (Active Comparator): Waitlist.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Tailored Internet-administrated CBT-Treatment — This intervention contains 6-8 text-based self-help modules in which 4 modules are fixed (the first three and the last) and the rest are "prescribed following the diagnostic telephone interview. These modules contain material on panic disorder, social phobia, stress management, assertiveness training, concentration, relaxation among other things.
  Arms: Tailored Internet-delivered CBT
Behavioral: Waitlist — Passive waitlist during 8-10 weeks.
  Arms: Waitlist

SUMMARY:
The purpose of this study is to determine whether tailored internet-administrated CBT is a feasible approach in the treatment of panic symptoms and comorbid anxiety and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-30 years old or 31-46 years old
* Have reoccurring panic attacks

Exclusion Criteria:

* Suicide prone
* Alcohol addiction
* PTSD
* OCD
* Ongoing psychological treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Panic Disorder Severity Scale (PDSS) | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in panic symptoms two weeks post treatment, at six months and at 12 months post treatment.

SECONDARY OUTCOMES:
Clinical Outcome in Routine Evaluation - Outcome Measure (CORE-OM) | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety and depressive symptoms two weeks post treatment, at six months and at 12 months post treatment.
Beck Anxiety Inventory (BAI) | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.
Montgomery Åsberg Depression Rating Scale-Self Rated (MADRS-S) | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in depressive symptoms two weeks post treatment, at six months and at 12 months post treatment.
Quality of Life Inventory (QOLI) | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in quality of life statements two weeks post treatment, at six months and at 12 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Department of Behavioral Sciences and Learning, Linköping University

REFERENCES:
- [Derived] Silfvernagel K, Carlbring P, Kabo J, Edstrom S, Eriksson J, Manson L, Andersson G. Individually tailored internet-based treatment for young adults and adults with panic attacks: randomized controlled trial. J Med Internet Res. 2012 Jun 26;14(3):e65. doi: 10.2196/jmir.1853. PMID 22732098